CLINICAL TRIAL: NCT00978276
Title: Concordance Study for Over Expression Level of Antibodies Within Breast Tissues
Brief Title: Immunohistochemical (IHC) Scoring for Receptors Expression in Breast Tissues
Status: Withdrawn | Type: Observational
Why Stopped: Personal changes in the company
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Tsafrir Kolatt, Applied Spectral Imaging Ltd.
Other Study IDs: ASI-IHC
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: Receptors; Immunohistochemistry; Breast; Over expression of Hormone receptors in carcinoma of the breast sues
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin embedded tissue sections of the breast
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is the identification and classification of human tissues and cytology specimens and elements therein.

Computer aided technology to assist the pathologists to identify, quantify, characterize and report their findings with regards to one or more diagnoses they should perform. In particular and for example: the scoring of the number of elements and their protein (antibody) expression level within a paraffin embedded tissue section.

ELIGIBILITY:
Inclusion Criteria:

* Well stained paraffin embedded tissue specimens

Exclusion Criteria:

* Fade away slides

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The breast samples were taken from female patients after tru cut biopsies, lumpectomies or mastectomies. Paraffin embedded blocks were prepared from the specimens out of which sections were stained immunohistochemically with the Vision Bio Systems mouse monoclonal antibodies for Estrogen Receptor (NCL-ER-6F11) and Progesterone Receptor (NCL-PGR-312). All stages were performed under the routine procedure of the hospital laboratory.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-05